CLINICAL TRIAL: NCT00275327
Title: Mechanisms of Resistance and Molecular Epidemiology of Commonly Encountered Multi-Resistant Bacteria
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Responsible Party: Sponsor
Other Study IDs: IRB# 0510165
Record Dates: First submitted 2006-01-09; First posted 2006-01-11 (Estimated); Last update posted 2015-12-17 (Estimated); Status verified 2015-12

CONDITIONS: Bacterial Infection
Keywords: antibiotics
MeSH Terms: conditions — Bacterial Infections

STUDY DESIGN:
Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — No genetic testing will be performed on any of the samples being obtained. The biologic samples will be under the control of the principal investigator of this research project. To protect confidentiality, all personal identifiers (i.e., name, social security number, and birth date) will be removed (de-identified) and replaced with a specific code number. The information linking these code numbers to the corresponding subjects' identities will be kept in a separate, secure location. The investigators on this study will keep the samples indefinitely. If a subject withdraws and provides the request in writing, samples collected and not already processed will be destroyed. All samples will be kept in the investigator's laboratory located in Scaife Hall, Room 812, 3550 Terrace Street.
Oversight: Data Monitoring Committee: Yes

SUMMARY:
o determine if extended-spectrum beta-lactamases, plasmid-mediated AmpC beta-lactamases, carbapenemases, chromosomal mutations in ribosomal RNA or other mechanisms of resistance account for antibiotic resistance in commonly encountered Gram negative and Gram positive bacteria at UPMC. Also to determine the molecular epidemiology and in vitro susceptibility of multiply resistant organisms at UPMC and to relate this to antibiotic use in the institution.

DETAILED DESCRIPTION:
The following variables will be followed: time and location of positive cultures, underlying diseases and severity of illness, recent immunomodulative therapies, physical exam findings, laboratory and radiographical data, antimicrobial usage of onset of infection, microbiological data and resistance patterns, choice of antibiotics once organism identified, suspected source of infection, bacteriological outcomes, laboratory results, demographic information, medications, clinical outcome gender, height, weight, ethnicity, and past medical history. The following variables will be followed: time and location of positive cultures, underlying diseases and severity of illness, recent immunomodulative therapies, physical exam findings, laboratory and radiographical data, antimicrobial usage of onset of infection, microbiological data and resistance patterns, choice of antibiotics once organism identified, suspected source of infection, bacteriological outcomes, laboratory results, demographic information, medications, clinical outcome gender, height, weight, ethnicity, and past medical history. The bacteria in the patient's cultures will be subcultured (after the diagnosis has been obtained since the microbiology lab would otherwise destroy the culture) and provided to the honest broker who will deidentify the specimen and link it to the medical information collected (which will also be deidentified by the honest broker). Patient data will be entered into a database by the honest brokers using an excel program for electronic data capture and reporting system. The honest brokers will have access to the database to ensure data integrity and perform data analyses. In addition, the Honest Broker will obtain information from the medical record as well as information about the specimens. The research team will have access to the database that is deidentified. The following evaluation will be performed on the bacteria. The minimal inhibitory concentration of the antibiotic used in treatment will be performed by the E-Test method (AB Biodisk, Solna, Sweden). Specific mechanisms of antimicrobial resistance will be studied with emphasis on the molecular mechanisms of antibiotic resistance such as production of beta-lactamases. This evaluation will be performed by analytical isoelectric focusing techniques as well as PCR and gene sequencing analysis to determine genes encoding beta-lactamases. Biologic samples will be under the control of the principal investigator of this research project. All samples provided to the investigators are deidentified by the honest broker and will be coded with numbers. The information linking these code numbers to the corresponding subjects' identities will be kept in a separate, secure location that only the honest broker has access to. The investigators on this study will keep the samples indefinitely. Samples will be kept in the investigator's laboratory located in Scaife Hall, room 812, 3500 Terrace Street. At no time will the research investigators have access to any patient identifiers.

ELIGIBILITY:
Inclusion Criteria:

* bacteria resistant to commonly used antibiotics

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: isolates
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2006-01; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yohei Doi, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania, United States